CLINICAL TRIAL: NCT07394764
Title: Development of a Physical Activity and Exercise Program Model for Children's Psychosocial Health and Physical Fitness Levels in Disasters: A Container City Example in the Earthquake Zone
Brief Title: Exercise Intervention in Children Living in a Container City
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Filiz Özdemir, ASSOCIATE PROFESSOR DR., Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Inonu; 323S479 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: This Study Focuses on Children Affected by the Earthquake
Keywords: Disaster; physical activity; exercise; psychosocial health; physical fitness; container city
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Warm-Up Exercise; Cool-Down Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): This study plans for a 12-week exercise training program, implemented three days a week. Children and families planned for inclusion in the experimental group will receive training on the importance of physical activity, the risks of a sedentary lifestyle, and daily physical activity recommendations, along with brochures. A daily logbook will be kept, and each child's information will be recorded in detail. On designated days, 60-minute sessions will be conducted, combining aerobic and strength training with play-based recreational activities. Each session will consist of 30 minutes of aerobic exercise and 10 minutes of strength training. Warm-up, cool-down, and relaxation exercises will be provided at the beginning and end of each session.
  Interventions: Other: Exercise
- control group (No Intervention): Children in the control group will not receive any exercise training. This group will continue with their routine lives.

INTERVENTIONS:
Other: Exercise — 934 Children and families planned for inclusion in the experimental group will receive training on the importance of physical activity, the risks of a sedentary lifestyle, and daily physical activity recommendations, along with brochures. On designated days, 60-minute sessions will be conducted, combining aerobic and strength training with play-based recreational activities. Each session will consist of 30 minutes of aerobic exercise and 10 minutes of strength training. Warm-up, cool-down, and relaxation exercises will be provided at the beginning and end of each session. The exercise program will be individualized according to the FITTE principle. The FITTE principle involves creating an individual exercise prescription based on the steps (Frequency, Intensity, Type, Time, Enjoy).
  Other Names: warm-up exercise; aerobic exercise; strengthening exercise; relaxation exercises; cool-down exercise
  Arms: intervention group

SUMMARY:
Disasters are natural events that deeply affect human life and can lead to psychosocial problems. Major disasters such as earthquakes can also jeopardize children's health both physically and psychologically. Children may suffer neurological, orthopedic, and traumatic injuries, in addition to the trauma of entrapment, displacement, loss of loved ones, and the upheaval of their daily lives during such events. These traumatic experiences can induce mental health issues like anxiety and depression, as well as physical symptoms such as fatigue, sleep disturbances, energy deficiency, and concentration loss. Post-earthquake, there is an observed increase in lifestyle-related illnesses, with individuals in temporary accommodations experiencing reduced physical activity levels, heightening the risk of these conditions.

Although the health benefits of physical activity are well-documented, the aftermath of earthquakes can deter motivation for exercise due to housing and environmental challenges. Consequently, specialized strategies are advocated to promote physical activity and enhance individual self-confidence. The unique value of this research project is to explore the psychosocial advantages of physical activity in post-earthquake scenarios for children, emphasize the role of physiotherapists, and develop a model for countries in seismic zones, including our own. The proposal aims to protect and improve the health of children aged 6-10 residing in post-earthquake container cities through a designated station to increase physical activity.

This project proposes:

* The creation of a physical activity unit in our country's frequently erected temporary housing for disaster victims, which typically lacks facilities to support children's physical and psychosocial health. This unit is envisioned to serve as a model.
* The design of a motivating and suitable environmental setting within the proposed unit for children whose activity opportunities have been curtailed post-earthquake.
* The role of the unit in safeguarding and enhancing the health of children following a disaster.
* The inclusion of child-specific, programmed, and engaging activities within the unit to boost children's physical performance and enable them to spend their free time productively.

The research will be conducted in a container city established in Malatya's center following the earthquakes on February 6, 2023, which houses a significant density of children aged 6-10. The study will involve more children than the number determined by power analysis, divided randomly into experimental and control groups. The experimental group will participate in a program at a physical activity and exercise station established in the container city, under the guidance of physiotherapists. The program will feature diverse and individualized exercise models, with suitable environmental modifications and equipment provided at the exercise station to facilitate age-appropriate activities. A 12-week training program is planned for the experimental group, while the control group will not receive any training. Outcome measures will include assessments of the children's psychosocial health and physical fitness, conducted at the program's inception, the 12th week, and subsequently the 24th week.

Upon completion, the project is expected to:

* Enable children in temporary housing to spend their time beneficially through scientifically guided training programs, thereby assuming a protective role.
* Serve as an exemplary model for intervention programs catering to the diverse needs of children requiring physical activity and exercise in temporary housing.
* Prepare the ground for integrating physical activity and exercise station units in future temporary housing established in the wake of natural disasters, thus contributing to disaster management.
* Ensure the stations are cost-effective, accessible, and financially efficient.

ELIGIBILITY:
Inclusion Criteria:

* Being between 6-10 years old
* Permanently residing in a container city
* Family and child consent to participate in the study

Exclusion Criteria:

* Presence of a metabolic disease (celiac disease, diabetes, thyroid disorders, obesity, etc.)
* Presence of a neuromuscular disease (cerebral palsy, muscle diseases, spina bifida, etc.)
* Presence of a cardiopulmonary disease (congenital heart diseases, asthma, cystic fibrosis, etc.)
* BMI percentile value between <5 and >99
* History of psychiatric diagnosis and treatment according to DSM-5 criteria
* Having a neurodevelopmental disorder (autism, mental retardation, etc.)
* Having a diagnosis of schizophrenia and bipolar disorder, etc.
* Children who are on chronic medication for any medical reason
* Having hearing, visual, or orthopedic impairment

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
physical fitness | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  The physical fitness levels of the participating children will be assessed using the European Fitness Tests (EuroFIT) battery.
psycosocial health-quality of life | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  Developed in 1999, Pediatric Scale Quality of Life (PEDSQL) scale is designed to assess General Health-Related Quality of Life in children and adolescents aged 2-18 years. It includes both a parent-report form and a self-report form completed by children and adolescents. The scale consists of 23 items and yields scores in three domains: the Total Scale Score (TSS), the Total Physical Health Score (PHHS), and the Total Psychosocial Health Score (PSHS). The PSHS is derived from items assessing emotional, social, and school functioning.
psychosocial health-Strengths and Difficulties Questionnaire | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  Another instrument used to screen for mental health problems in children and adolescents is the Strengths and Difficulties Questionnaire (SDQ), developed by Robert Goodman in 1997. The SDQ is designed for use with children and adolescents aged 4-16 years. It consists of 25 items and serves as a screening tool for the early identification of psychological difficulties and a range of behavioral and emotional problems in children.
psychosocial health - Depression Scale | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  The DSM-5 Level 2 Depression Scale - Parent Form assesses depressive symptoms experienced by children over the past 7 days. The scale includes a parent-report form applicable to children aged 6-17 years and a self-report form completed by adolescents aged 11-17 years. In the present study, the parent-report form will be used. The parent form consists of 11 items.
psychosocial health - Anxiety Scale | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  The DSM-5 Level 2 Anxiety Scale - Parent Form is designed for use in the initial assessment and treatment monitoring of children and adolescents with anxiety disorders. The scale evaluates the severity of anxiety symptoms experienced by children and adolescents during the past 7 days, with higher scores indicating greater anxiety severity.
  The instrument includes a 10-item parent-report form completed by a parent or guardian for children aged 6-17 years, as well as a 13-item self-report form completed by adolescents aged 11-17 years. In the present study, the parent-report form will be used.
psychosocial health-Post-Traumatic Stress Scale | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  The Childhood Post-Traumatic Stress Disorder Scale (PEDS), developed by Saylor in 1999, is designed to assess behavioral symptoms associated with Post-Traumatic Stress Disorder in children aged 2-10 years. The scale consists of 21 items and is completed by caregivers. Items are rated on a Likert-type scale, yielding a total score ranging from 0 to 84, with higher scores indicating greater severity of post-traumatic stress symptoms.
psychosocial health - Psychiatric Condition Assessment | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  The K-SADS-PL, developed by Kaufman and colleagues in 1997 to identify psychiatric conditions in children and adolescents aged 6-18 years, is a semi-structured psychiatric interview that was revised in 2016 in accordance with DSM-5 diagnostic criteria. The interview consists of several stages.
  The first section collects information on sociodemographic characteristics, presenting complaints, developmental history, health status, and functioning in school and home environments. The second section includes screening questions that assess both past and current psychiatric symptoms, with current symptoms referring to those present within the past two months. The third section consists of assessment and observational findings used to confirm DSM-5 diagnoses.
  Information obtained from each source is scored separately and subsequently integrated with the clinician's observations to reach the final diagnostic evaluation.
Sociodemographic and General Physical Examination Characteristics | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention
  The sociodemographic characteristics of the participating children-including age, sex, school and grade level, family structure, number of siblings, family socioeconomic status, and parental education level-will be assessed using a structured questionnaire. In addition, information related to the earthquake experience (such as losses, school-based support, and peer support) will also be collected.
  General physical examination findings, including body weight, height, and blood pressure, will be measured and recorded.
psychosocial health - Stress Axis Activities | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  Salivary cortisol levels will be measured to determine the stress hormone profiles of the participants. To minimize the effects of confounding factors, cortisol sampling will be conducted between 09:00 and 11:00 a.m. for all participants, as salivary cortisol levels are known to become relatively stabilized after 09:00 a.m.
  The primary parameter to be evaluated is not the absolute cortisol level itself, but rather the change in state anxiety levels and salivary cortisol concentrations before and after the intervention.
Physical Activity Level | Baseline, at the end of the 12-week intervention, and at the end of the 24-week intervention.
  The Children's Physical Activity Questionnaire will be used to assess the physical activity levels of the participants. This questionnaire was originally developed in Canada as the Physical Activity Questionnaire for Older Children (PAQ-C).

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves children living in a disaster-affected area, and sharing de-identified individual-level data could pose potential risks related to participant privacy and confidentiality. In addition, informed consent does not include provisions for sharing IPD with external researchers.